CLINICAL TRIAL: NCT05159336
Title: Intervention Treatment of Auditory Hallucination by Transcranial Alternating Current Stimulation
Brief Title: Transcranial Alternating Current Stimulation (tACS) for Auditory Hallucinations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDYX20211101
Record Dates: First submitted 2021-11-10; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- schizophrenia patients with auditory hallucinations (Experimental): For schizophrenia patients with auditory hallucinations, tACS for implementation intervention
  Interventions: Device: tACS for auditory hallucinations via single arm

INTERVENTIONS:
Device: tACS for auditory hallucinations via single arm — a 20 weeks, weekly 40 minutes, 1mA, 10Hz-tACS protocol

SUMMARY:
Transcranial alternating current stimulation (tACS) can modulate and restore neural oscillations that are reduced in patients with psychiatric illnesses such as schizophrenia. Here, we performed a open-lable study of clinical trial in 30 schizophrenia patients with auditory hallucinations to show that tACS is effective for auditory hallucinations.

DETAILED DESCRIPTION:
Each week, the patient rested quietly with her eyes open while receiving alpha-frequency tACS for 40 minutes. Stimulation was delivered at 10 Hz with 1 mA zero-to-peak amplitude in-phase to the location 1 and the location 2 acquired by the MEG technique with 5*5 cm electrodes. A 5* 7 cm return electrode was centered on Cz. In total, 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia with auditory hallucinations was diagnosed by DSM-IV, AHRS >12, Take sufficient antipsychotics for at least 1 month.

Exclusion Criteria:

* current pregnancy, major medical illness affecting the central nervous system, significant neurologic disorders, intake of drugs including supplements like essential fatty acids that influence prostaglandins or niacin skin flush flash pathway metabolism, a history of suicide risk, or alcohol or drug abuse.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-28 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Auditory Hallucination Scale(the minimum is 0, maximum value is 47, and higher scores mean a worse outcome) | One month
  Reduction rate of AHRS scale

CONTACTS AND LOCATIONS:
Overall Officials: Yegang Hu, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Force RB, Riddle J, Jarskog LF, Frohlich F. A case study of the feasibility of weekly tACS for the treatment of auditory hallucinations in schizophrenia. Brain Stimul. 2021 Mar-Apr;14(2):361-363. doi: 10.1016/j.brs.2021.01.014. Epub 2021 Jan 27. No abstract available. PMID 33515747
- [Result] Ahn S, Mellin JM, Alagapan S, Alexander ML, Gilmore JH, Jarskog LF, Frohlich F. Targeting reduced neural oscillations in patients with schizophrenia by transcranial alternating current stimulation. Neuroimage. 2019 Feb 1;186:126-136. doi: 10.1016/j.neuroimage.2018.10.056. Epub 2018 Oct 24. PMID 30367952